CLINICAL TRIAL: NCT04620603
Title: Low-Dose-Rate Brachytherapy Combined With Immune Checkpoint Inhibition in Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE6620
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Cutaneous Malignant Melanoma; Renal Cell Cancer; Urothelial Cancer of Renal Pelvis
Keywords: Brachytherapy
MeSH Terms: conditions — Melanoma, Cutaneous Malignant; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- LDR + SOC Immunotherapy (Experimental): Participants will receive one treatment of brachytherapy on treatment day 1 (LDRD1). After a minimum of 7 days but no more than 30 days to allow antigenic release, participants will then begin immunotherapy treatment with SOC immunotherapy at the standard FDA-approved dose. Standard immunotherapy will be administered on D1 of every standard of care cycle (either 14, 21, 28, or 42 day cycle) at the standard dose. Participants can receive up to 1 year of SOC immunotherapy.
  Interventions: Radiation: Low Dose Rate Brachytherapy (LDR); Drug: Standard-of-Care Immunotherapy

INTERVENTIONS:
Radiation: Low Dose Rate Brachytherapy (LDR) — LDR on treatment day 1
Drug: Standard-of-Care Immunotherapy — Standard or care immunotherapy will be administered at the FDA approved dose via IV infusion.

SUMMARY:
This is a pilot study of combination low dose rate brachytherapy (LDR) added to standard of care (SOC) immunotherapy in stage III and IV melanoma, stage IV renal call cancer, and stage IV urothelial cancer.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of combining LDR with immune checkpoint inhibition in stage III and IV melanoma, stage IV renal call cancer, and stage IV urothelial cancer. This involves the addition of a treatment called brachytherapy to SOC immunotherapy. Brachytherapy is a form of radiation therapy where radioactive pellets are placed within a tumor to temporarily irradiate the tumor at a low level. This is the first time that this combination (immunotherapy and brachytherapy) has been used in humans.

The objectives of this study are to evaluate the effect of combining LDR with immunotherapy, determine safety and feasibility, generate a toxicity profile, evaluate response, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed unresectable stage III or stage IV cutaneous melanoma, stage IV renal cell cancer, and stage IV urothelial cancer.
* ECOG performance status 0-2.
* Have measurable disease per RECIST v1.1 or iRECIST. Refer to Appendix B
* Have the following clinical laboratory values:

  * Absolute neutrophil count (ANC) ≥ 1500/ μL
  * Hgb ≥ 9 g/dL
  * Platelet count ≥ 75, 000/ μL
  * Total bilirubin ≤ 1.5 x ULN (upper limit of normal)
  * AST and ALT ≤ 2x ULN
  * Serum Creatinine < 2x ULN
* Female participants who:

  * Are postmenopausal for at least 1 year before entering the screening visit, OR
  * Are surgically sterile, OR
  * Agree to practice true abstinence from heterosexual contact or agree to use effective contraception without interruption during the study therapy and 90 days after the last dose.
* Male participants who:

  * Are surgically sterile, OR
  * Agree to practice true abstinence from heterosexual contact or agree to use effective contraception without interruption during the study therapy and 90 days after the last dose.

Exclusion Criteria:

* Participants diagnosed with uveal melanoma
* Participants who have been treated with whole head radiation for brain metastases
* Invasive cancers not being treated on this trial (i.e. lymphoma that received systemic therapy) diagnosed < 3 years prior that required systemic treatment. This is intended to include a patient with melanoma who was diagnosed < 3 years prior to screening for this trial that has received antecedent systemic therapy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Prior anti-cancer therapy for melanoma, renal cell cancer, or urothelial cancer less than 14 days prior to first dose of study treatment.
* Pregnant or nursing females
* Unwilling or unable to follow protocol requirements.
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study treatment.
* Other active non-melanoma, non-renal cell, or non-urothelial metastatic cancers requiring systemic treatment.
* Participants currently receiving systemic corticosteroids doses over 15mg prednisone or equivalent.
* Participants with uncontrolled HIV or hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with tumor response assessed by Immunotherapy Response Evaluation Criteria in Solid Tumors (iRECIST) | 3 months after brachytherapy
  iRECIST was developed by the RECIST working group for the use of RECIST version 1.1 in cancer immunotherapy trials, to ensure consistent design and data collection.
  ORR is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on iRECIST or RECIST v1.1 at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on CT or MRI scans
Number of participants with tumor response assessed by Immunotherapy Response Evaluation Criteria in Solid Tumors (iRECIST) | 6 months after brachytherapy
  iRECIST was developed by the RECIST working group for the use of RECIST version 1.1 in cancer immunotherapy trials, to ensure consistent design and data collection.
  ORR is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on iRECIST or RECIST v1.1 at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on CT or MRI scans
Number of participants with tumor response assessed by Immunotherapy Response Evaluation Criteria in Solid Tumors (iRECIST) | 9 months after brachytherapy
  iRECIST was developed by the RECIST working group for the use of RECIST version 1.1 in cancer immunotherapy trials, to ensure consistent design and data collection.
  ORR is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on iRECIST or RECIST v1.1 at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on CT or MRI scans
Number of participants with tumor response assessed by Immunotherapy Response Evaluation Criteria in Solid Tumors (iRECIST) | 12 months after brachytherapy
  iRECIST was developed by the RECIST working group for the use of RECIST version 1.1 in cancer immunotherapy trials, to ensure consistent design and data collection.
  ORR is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on iRECIST or RECIST v1.1 at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on CT or MRI scans
Number of participants with tumor response assessed by RECIST v1.1 | 3 months after brachytherapy
  ORR is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on the Response Evaluation Criteria in Solid Tumors (iRECIST or RECIST v1.1) at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on CT or MRI scans
Number of participants with tumor response assessed by RECIST v1.1 | 6 months after brachytherapy
  ORR is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on iRECIST or RECIST v1.1 at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on CT or MRI scans
Number of participants with tumor response assessed by RECIST v1.1 | 9 months after brachytherapy
  ORR is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on iRECIST or RECIST v1.1 at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on CT or MRI scans
Number of participants with tumor response assessed by RECIST v1.1 | 12 months after brachytherapy
  ORR is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on iRECIST or RECIST v1.1 at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on CT or MRI scans

CONTACTS AND LOCATIONS:
Overall Officials: Jay Ciezki, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared but the study team is expecting to publish the data